CLINICAL TRIAL: NCT03839667
Title: Effect of Intermittent Intensive Diet Intervention and Enhanced Physical Activity on Glycemic Control in Patients With Newly Diagnosed Type 2 diabEtes (IDEATE)
Brief Title: Intensive Diet and Physical Activity on Diabetes
Acronym: IDEATE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Guang Ning, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ruijin-2018-174-2
Record Dates: First submitted 2019-01-06; First posted 2019-02-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Type2 Diabetes; Life Style

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intensive diet intervention group (Experimental): The participants will be instructed to restrict the total daily calorie intake to 800 kcal by receiving the very-low-calorie meal replacement formula for 2 consecutive days per week. They will be allowed to maintain their normal diet in the remaining 5 days, but need to restrict total intake to 2000 kcal per day.
  Interventions: Behavioral: intensive diet intervention
- Enhanced physical activity group (Experimental): the participants will take high-intensity exercise in accordance with High Intensity Interval Training (HIIT) prescriptions, with maximum heart rate and relative maximal oxygen uptake monitored. They will take both aerobic and resistance training exercise consecutively, and total training time will be expected to reach at least 150 minutes per week.
  Interventions: Behavioral: Enhanced physical activity intervention
- Standard education group (Experimental): the participants will receive no extra intervention but diabetes health education, which will be carried out in large classrooms, in groups, and over the telephone. The education is mainly consisted of instructions on healthy diet and exercise plans, prevention for acute and chronic complications and self-glycemic monitoring.
  Interventions: Behavioral: Standard education

INTERVENTIONS:
Behavioral: intensive diet intervention — the participants will be instructed to restrict the total daily calorie intake to 800 kcal by receiving the very-low-calorie meal replacement formula for 2 consecutive days per week. They will be allowed to maintain their normal diet in the remaining 5 days, but need to restrict total intake to 2000 kcal per day.
  Arms: intensive diet intervention group
Behavioral: Enhanced physical activity intervention — the participants will take high-intensity exercise in accordance with High Intensity Interval Training (HIIT) prescriptions, with maximum heart rate and relative maximal oxygen uptake monitored. They will take both aerobic and resistance training exercise consecutively, and total training time will be expected to reach at least 150 minutes per week.
  Arms: Enhanced physical activity group
Behavioral: Standard education — the participants will receive no extra intervention but diabetes health education, which will be carried out in large classrooms, in groups, and over the telephone. The education is mainly consisted of instructions on healthy diet and exercise plans, prevention for acute and chronic complications and self-glycemic monitoring.
  Arms: Standard education group

SUMMARY:
It is a multicenter, open-label, parallel-group, randomized controlled clinical trial, which is designed to enroll newly diagnosed type 2 diabetes patients with overweight or obesity. The patients are randomized to an intensive diet intervention (intermittent very-low -calorie diet), enhanced physical activity intervention (high-intensity interval training exercise prescription combined with resistance training) or standard education group (diabetes health education only, including lifestyle education and guidance) for 12 weeks. This trial will test the primary hypothesis of whether an intensive lifestyle treatment (diet or physical activity) is more effective than a standard education in glycemic control. The secondary hypotheses are to compare the intensive lifestyle treatment with a standard education on adipose distribution, metabolic parameters, metabolic molecules, Framingham Risk Scores, and quality of life, et al.

DETAILED DESCRIPTION:
The trial will recruit 324 patients from 2-3 hospitals within the China Diabetes Clinical Research Network. Eligible criteria include men and women aged 40-70 years; newly-diagnosed type 2 diabetes mellitus; BMI ≥25 kg/m2 and <40 kg/m2. Main exclusion criteria include known type 1 diabetes, usage of insulin; symptomatic cardiovascular diseases, and other serious illness. The proposed trial has 90% statistical power to detect an absolute 0.5% reduction of HbA1c changes between intensive intervention and standard education groups at a 2-sided significance level of 0.05. To achieve the proposed study objectives, we plan to perform the following specific aims:

1. Recruit 324 study participants who meet the eligibility criteria and randomly assign 108 to the intensive diet intervention group, 108 to the enhanced physical activity intervention group and 108 to the standard education group for 12 weeks;
2. Employ a study-wide strategy to encourage standard of care for all participants for the treatment of type 2 diabetes and other metabolic disorders;
3. Obtain clinical data on study outcomes for up to 12 months of follow-up among all trial participants;
4. Perform strict quality control procedures for intervention and data collection;
5. Conduct data analysis according to the intention-to-treat principle;
6. Disseminate the study findings to influence clinical practice and clinical guidelines.

The results will be analyzed to examine the pan-omics changes after the interventions and clarify their predictive benefits on the effects of the interventions.

After the 12-week intervention, participants will receive post-intervention follow-up visits at 24 weeks, 36 weeks, 48 weeks, and 5 years from the baseline enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 40-70 years;
2. Newly diagnosed type 2 diabetes

   * Duration of type 2 diabetes ≤ 2 years;
   * Antidiabetic treatment maintained for at least 6 weeks before recruitment;
3. 7.0%≤ HbA1c < 9.0%;
4. 25 Kg/m2 ≤ Body mass index (BMI) <40 Kg/m2;

Exclusion Criteria:

1. History consistent with type 1 diabetes;
2. Insulin treatment;
3. Severe cardiovascular disease:

   * current angina
   * myocardial infarction within last six months
   * heart failure
   * symptomatic periphery vascular disease
4. Uncontrolled hypertension: systolic blood pressure > 180 mmHg or diastolic blood pressure > 100 mmHg;
5. Myocardial ischemia indicated by resting ECG;
6. Foot ulcers, peripheral neuropathy or skeletal disorders;
7. Taking high intensity exercise more than 75 minutes or moderate intensity exercise more than 150 minutes per week during the screening phase
8. Average weekly alcohol intake >140 grams for men and >70 grams for women;
9. ALT or AST levels more than twice the upper limit of the normal range or active liver diseases;
10. eGFR <60 ml/min/1.73 m2, or serum creatinine >1.5 mg/dl for men or 1.3mg/dl for women; or Proteinuria
11. Malignant tumor in active-stage, or in remission stage but less than 5 years from the most recent treatment
12. Hemoglobin concentration <130 g/l for men or <120 g/l for women;
13. Past or present confirmed psychiatric illness or drug dependence;
14. History of food allergies;
15. Surgical history of digestive system;
16. Currently taking medications known to affect weight (e.g. anti thyroid drugs, glucocorticoids);
17. Known to have weight-affecting diseases (e.g. malabsorption, functional bowel disease, uncontrolled low sodium/hyperthyroidism, eating disorders);
18. Known to have metabolism-affecting diseases;
19. Known to have infectious diseases within last month;
20. Possible consumption of food or drugs affecting glucose homeostasis or gut microbiota within the last three months;
21. Other acute diseases supported by clinical evidence which may contradict to the interventions;
22. Pregnancy, currently trying to become pregnant, or of child-bearing potential and not using birth control;
23. Currently participating in another intervention study;
24. Failure to obtain informed consent from participant;
25. Any factors judged by the clinic team to be likely to limit adherence to interventions;
26. Any other medical condition judged by the clinic team not eligible for the trial.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2026-03-21 (Estimated)

PRIMARY OUTCOMES:
change in HbA1C level (%) | 12 weeks

SECONDARY OUTCOMES:
change in HbA1C level (%) | From enrollment to the end of follow-up at 5 years
proportion of reversal of diabetes | From enrollment to the end of follow-up at 5 years
reduction in the dosage of hypoglycemic drugs | From enrollment to the end of follow-up at 5 years
change in insulin sensitivity | From enrollment to the end of follow-up at 5 years
  Quantify by HOMA score, which is calculated multiplying fasting plasma insulin (FPI, mIU/L) by fasting plasma glucose (FPG, mmol/L), then dividing by the constant 22.5, i.e. HOMA-IR = (FPI×FPG)/22.5.
change in islet β-cell function | From enrollment to the end of follow-up at 5 years
  Quantify by HOMA score, which is calculated with fasting plasma insulin (FPI, mIU/L) and fasting plasma glucose (FPG, mmol/L), i.e. HOMA-β = 20*FPI/(FPG-3.5).
change in liver steatosis quantified by MRI-PDFF (percentage) | From enrollment to the end of follow-up at 5 years
change in body mass index (BMI) | From enrollment to the end of follow-up at 5 years
  Body weight (kg) and height (m) will be combined to report BMI in kg/m^2
change in visceral fat (cm^2) | From enrollment to the end of follow-up at 5 years
change in serum fetuin-A concentration (μg/mL) | From enrollment to the end of follow-up at 5 years
change in serum GREM2 concentration (pg/ml) | From enrollment to the end of follow-up at 5 years
change in serum Caspase-cleaved Keratin 1 concentration (U/L) | From enrollment to the end of follow-up at 5 years
changes in serum FGF21 concentration (pg/ml) | From enrollment to the end of follow-up at 5 years
changes in overall gut microbiota profile | From enrollment to the end of follow-up at 5 years
  change in gut microbiota composition and proportion of specific gut flora.
depression | From enrollment to the end of follow-up at 5 years
  Evaluated with PHQ-9 scores. The PHQ is 59-question instrument, referring to the level of interest in doing things, feeling down or depressed, difficulty with sleeping, energy levels, eating habits, self-perception, ability to concentrate, speed of functioning and thoughts of suicide. Responses range from "0" (Not at all) to "3" (nearly every day).The total sum of the responses suggests varying levels of depression. Scores range from 0 to 27. In general, a total of 10 or above is suggestive of the presence of depression.
health related quality of life | From enrollment to the end of follow-up at 5 years
  Evaluated with HQoL scales such as Short Form 12 Health Survey Questionnaire
cardiovascular risk | From enrollment to the end of follow-up at 5 years
  Evaluated with Framingham Risk Scores. Individuals with low risk have 10% or less CHD risk at 10 years, with intermediate risk 10-20%, and with high risk 20% or more.

CONTACTS AND LOCATIONS:
Overall Officials: Guang Ning, MD, PhD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Ruijin hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided